CLINICAL TRIAL: NCT01490528
Title: Durability and Tolerability of Infliximab in Pediatric Inflammatory Bowel Disease Patients: A 10 Year Single Center Experience
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Marla Dubinsky, Director Pediatric IBd Center, Cedars-Sinai Medical Center
Other Study IDs: REMICADEIBD4008
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Pediatric Inflammatory Bowel Disease
Keywords: Pediatric IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is little data published on the long term durability of infliximab in pediatric patients. In particular a focus on durable remission, frequency of dose/frequency change and switch within class. Moreover 10 years of safety experience is rarely reported in children.

The overall objective is to evaluate the persistence of infliximab as well as dosing strategies in pediatric inflammatory bowel disease (IBD) patients and safety of infliximab Regarding persistence of infliximab the investigators will be focusing on the proportion of patients who continue to have a durable response or remission to infliximab.

The investigators will be assessing this by measuring the frequency of dose escalation, proportion of patients needing frequency change and proportion of patients switched to adalimumab or certolizumab.

Safety outcomes will focus on frequency of malignancies, infections and immunogenecity

ELIGIBILITY:
Inclusion Criteria:

* All individuals who received at least 2 doses of infliximab before the age of 16 at the pediatric IBD Center at Cedars Sinai Medical Center for the treatment of Crohn's disease or ulcerative colitis Able to give consent

Exclusion Criteria:

* not exposed to infliximab

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All individuals who received at least 2 doses of infliximab before the age of 16 at the pediatric IBD Center at Cedars Sinai Medical Center for the treatment of Crohn's disease or ulcerative colitis Able to give consent
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01

PRIMARY OUTCOMES:
Frequency of patients with a sustained durable remision and frequency of serious infections and malignancies in children exposed to infliximab | 10 years

SECONDARY OUTCOMES:
Frequency of concomitant immunomodulator use in children on infliximab | 10 years
Frequency of anti-drug antibodies in patients on and off comcomitant immunomodulators | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Marla Dubinsky, Principal Investigator — Cedar Sinai Medical Center